CLINICAL TRIAL: NCT01509963
Title: Prospective Evaluation of the Reliability of the Combined Use of Two Models to Predict Non-sentinel Lymph Node Status in Breast Cancer Patients With Metastatic Sentinel Lymph Nodes: the MSKCC Nomogram and the Tenon Score.
Brief Title: The Memorial Sloan-Kettering Cancer Center (MSKCC
Acronym: NOTEGS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI 10073; AOM 10220 (Other: Assistance Publique - Hôpitaux de Paris)
Record Dates: First submitted 2011-12-06; First posted 2012-01-13 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Breast Cancer
Keywords: MSKCC nomogram; Tenon score; metastatic SN; low risk of metastatic non-SN; additional ALND
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients candidates for the SN procedure: The study will focus on patients candidates for the SN procedure as recommended by Saint-Paul de VENCE initially in 2005 but modified in 2009.
  Interventions: Other: no intervention : measure of score

INTERVENTIONS:
Other: no intervention : measure of score — To provide probability of non sentinel lymph node metastasis in case of metastatic lymph node according to MSKCC nomogram and Tenon score.

SUMMARY:
The purpose of this study is to prospectively evaluate the combined use of the MSKCC nomogram (Memorial Sloan-Kettering Cancer Center) and Tenon score to select, in patients with metastatic sentinel lymph node (SN), those at low risk of metastatic non-SN in whom additional axillary lymph node dissection (ALND) could be avoided.

DETAILED DESCRIPTION:
EXPERIMENTAL PLAN AND COURSE OF STUDY This is a prospective non-randomized non-interventional multicenter study including the respect of a quality charter and involving a prospective registration of clinical and histological data to test the hypothesis of a proportion of false negative rate (=rate of metastatic SN) of 5% +/- 5% within the population at low risk by the combined use of the MSKCC nomogram and Tenon score. No modification therapy will be conducted because the scores will not be provided to operators.

6.1 Conduct of the study 6.1.1 Before and during surgery Every surgeon agreeing to participate in the study - and thus to respect the quality charter - will make the inclusion of his eligible patients with an e-CRF which will generate automatically a number of anonymity. A form of inclusion specifying the number of anonymity of the patient, the initials of the name and the first name as well as the date of birth of the patient will be send back by e-mail by the study coordinator and clinical study technician (CST) of the URC-Est. The surgeon will have at his disposal 60 boards of labels of anonymity elaborated by the CST of the URC-Est corresponding to 30 patients (2 boards of labels by patient). The resupplying of labels will be managed by the CST.

A label will contain i) the number of anonymity, ii) the address and phone number of the surgeon, iii) the address and phone number of the pathology laboratory, iv) the address and phone number of the study coordinator including fax number where pathological results should be send.

During the first intervention, the surgeon will send the histological specimen (i.e. lumpectomy or mastectomy, SN, and possibly non-SN in case the ALND is completed during the first surgical procedure with a board of labels of anonymity.

In case of additional surgical procedure to complete ALND, the histological specimen (i.e. non-SN) will be sent to the pathology laboratory with the second board of label of anonymity corresponding to this patient.

The laboratory of pathology will have to label with anonymity labels all histological reports that should be sent to the study coordinator. To eventually calculate combined prediction (MSKCC nomogram and Tenon score) and ensure respect of the quality charter, specific data must appear in the pathology report:

* Clinical information: age of the patient, the location of the primitive tumor (upper outer quadrant, SUPERO-medial, INFERO-lateral, INFERO-internal retroareolar or other), palpable tumor or not, the results of histological or cytological diagnosis performed preoperatively.
* Regarding the number of lumpectomy: size of invasive cancer (largest diameter), histologic type, associated intra ductal carcinoma (type and percentage), existence of vascular or lymphatic emboli, estrogen receptor status, progesterone receptor status, HER-2-neu status, SCAFF and Bloom-Richardson grade or equivalent, if realized, the level of expression of antigen Ki 67; regarding sentinel lymph nodes: number of SN harvested ; for each metastatic SN: type of metastasis: macrometastasis, micrometastasis, isolated cells, method of intraoperative diagnosis of metastasis (if performed): frozen section, cytology, RT-PCR. Final pathologic exam: routine H&E, serial sectioning H&E, IHC. Regarding non-sentinel lymph nodes: number of non-SN
* number of metastatic non-SN, postoperative TNM. 6.1.2 Collection of histological results from the pathology laboratories The study data will be informed through pathology reports. Ten weeks after receiving the e-CRF, the CST of the URC-EST under the responsibility of the study coordinator will contact the pathology laboratory. The latter will label with anonymity labels all histology reports corresponding to the first and possibly, if an additional ALND has further been done, and will fax reports to the study coordinator(fax number on the label).

6.2 Procedure to calculate the risk of non-SN involvement A calculation of the probability of metastatic non-SN using the MSKCC nomogram and the the Tenon score will be performed for all patients. Calculations will be implemented under the responsibility of coordinating doctor.

The result of these calculations will not be communicated to surgeons. 6.2.1 Calculating the score of Tenon

* Variable 1: Existence of macrometastasis in a non-SN: if macrometastases, 2 points are assigned, 0 otherwise.
* Variable 2: histological size of invasive tumor: 3 points if the tumor is greater than 20 mm, 1.5 points if the size is in 10 and 20 mm and 0 points if less than 10 mm.
* Variable 3: Ratio between the number of metastatic SN (whatever the type of metastasis (macrometastasis, micrometastasis or isolated tumor cells)) and the number of SN harvested: 2 points if the ratio is 1; 1 point if between 0.5 and 1, and 0 points if less than 0.5.

The scores for the 3 variables are then added together to calculate the score of Tenon.

6.2.2 Calculation of risk by the MSKCC nomogram This calculation involves 8 variables: 1) histological type associated with SBR grade (infiltrating ductal carcinoma grade 1, grade 2, grade 3 and invasive lobular carcinoma (ILC)), 2) the existence of a LYMPHO-vascular invasion (LVI) (yes, no), 3) the multifocal nature of the tumor (yes, no), 4) status of estrogen receptor (present, absent), 4) the number of non-metastatic SN (0 to 14), 5) the number of metastatic SN (from 1 to 7), 6) the size of the tumor (from 0 to 9 cm), 7) method of detecting metastases in the SN. For the latter, there are 2 different situations: when using the technique CRYOCONGELATION, 4 items were proposed (CRYOCONGELATION analysis, analysis by H&E : routine H&E and serial sectioning H&E, and IHC), and in the absence of use of technology by cryocongelation only 3 items were proposed (analysis by H&E : routine H&E and serial sectioning H&E, and IHC).

1. The calculation must be done using the calculator developed by the authors and easily accessible on the website http://www.mskcc.org/MSKCC/htlm/5794.cfm.

   * First Row "Performed Frozen Section. The item must be checked if the pathologist has performed frozen section intra-operatively. Otherwise, the item must not be checked.
   * Second line "Pathological size (cm)" must refer the histological size of the largest tumor diameter in centimeters.
   * Third line "Tumor type and grade": you must select the corresponding item from the 4 items offered: ductal I (for infiltrating ductal carcinoma (TCC) grade 1), ductal II (for TCC grade 2), ductal III (for TCC grade 3) and lobular (for infiltrating lobular carcinoma).
   * Fourth line "Number of Positive Sentinel Lymph Nodes" must report the number of metastatic SN, whatever the type of flooding (by macrometastasis a micrometastasis or isolated cells).
   * Fifth line "SN Method of Detection": you must select the item. Two scenarios:

     1. In the first line item "Frozen Section Performed" was checked: 4 item are then offered: Frozen (if the metastasis was diagnosed at the frozen section). However, this scenario can not produce it because in this case, the patient has received ALND in the same operation as the procedure of SN; Routine (if the metastasis was diagnosed by analyzing routine H&E), Serial (if the metastasis was diagnosed after serial sectioning in H&E), IHC (if the metastasis was diagnosed by IHC)
     2. the first line item "Frozen Section Performed" was not checked: 3 item are then proposed: Routine (if the metastasis was diagnosed by analyzing routine H&E), Serial (if the metastasis was diagnosed after serial sectioning in H&E), IHC (if the metastasis was diagnosed by IHC).
   * Sixth row "Number of Negative Sentinel Lymph Nodes': the number of non-metastatic SN.
   * Seventh row "Lymphovascular Invasion." The item must be checked in case of lymphatic or vascular emboli.
   * Eighth row "Multifocality. The item must be checked in case of multifocality.
   * Ninth Line "Estrogen Receptor Positive". The item must be checked if the tumor estrogen receptors.
2. The use of the nomogram (defined as the graphical representation of the model) is not recommended because the calculation is less precise than the web interface.

6.2.3 Risk calculation combining the MSKCC nomogram and the Tenon score

* Group at low risk of metastatic non-SN: probability with the MSKCC nomogram of ≤ 10% and a score of Tenon ≤ 3.5.
* Group at risk of metastatic non-SN: probability with the MSKCC nomogram of > 10% and/or Tenon score > 3.5.

6.3 Monitoring of patients included in the study The study evaluates the combined use of two predictors at baseline. It does not require monitoring. However, all patients will be monitored regularly for any breast cancer and adjuvant treatment of breast cancer will remain unchanged by this study.

6.4 Total time of research The recruitment and the opening of study centers is planned over a period of 6 months. Inclusion of patients is planned over a period of 18 months. The total duration of the study is 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old with invasive breast cancer with an indication of SN procedure as recommended by Saint-Paul de VENCE in 2005 amended in 2009
* T1-2 breast cancer
* Patients having social security coverage.

Exclusion Criteria:

* Patient under the age of 18.
* Patient who had neoadjuvant chemotherapy.
* Patient who had had radiotherapy to the ipsilateral axilla or breast.
* Pregnant patient.
* Patients who do not speak French.
* Patients refusing to participate in the study.
* Simultaneous participation in another research period of exclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will focus on patients candidates for the SN procedure as recommended by Saint-Paul de Vence initially in 2005 but modified in 2009.
Sampling Method: Non-Probability Sample
Enrollment: 3194 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
False negative rate in patients with both a ≤ 10% probability of metastatic non-SN with the MSKCC nomogram and a Tenon score ≤ 3.5 (i.e. low risk): proportion of patients with metastatic non-SN at additional ALND. | after the surgery

SECONDARY OUTCOMES:
To determine the impact on the reliability of the combined predictor of frozen section examination in light of his achievement or not, and its sensitivity. | after the surgery
To allow, because of the large number of patients to include in the study, the diffusion of a charter of quality for the SN procedure. | after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Roman Rouzier, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Gynécologie Obstétrique et Médecine de la Reproduction Hôpital Tenon, 4 rue de la Chine, Paris, France